CLINICAL TRIAL: NCT02910141
Title: Individual Patient Data Meta-analysis of Randomised Controlled Trials Comparing Glycaemic Control During Continuous Subcutaneous Insulin Infusion vs. Multiple Daily Insulin Injections in Type 2 Diabetes Mellitus
Brief Title: Individual Patient Data Meta-analysis of CSII vs. MDI in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: University of Leicester (Other); University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Professor John Pickup, Emeritus Professor of Diabetes and Metabolism, King's College London
Other Study IDs: IPDMetaT2
Record Dates: First submitted 2016-09-12; First posted 2016-09-21 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Continuous subcutaneous insulin infusion; Meta-analysis; Insulin pump therapy; Multiple daily insulin injections
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CSII (subcutaneous insulin infusion): People with Type 2 diabetes treated by continuous subcutaneous insulin infusion (CSII)
  Interventions: Device: Continuous subcutaneous insulin infusion
- MDI (multiple daily insulin injections): People with type 2 diabetes treated by multiple daily insulin injections

INTERVENTIONS:
Device: Continuous subcutaneous insulin infusion — Infusion of short-acting insulin from a portable pump
  Other Names: Insulin pump therapy
  Groups: CSII (subcutaneous insulin infusion)

SUMMARY:
This study aims to compare glycaemic control during continuous subcutaneous insulin fusion (CSII, insulin pump therapy) and multiple daily insulin injections in type 2 diabetes and to identify patient-level characteristics that predict the best improvement in control and any change in insulin dose or other outcome.

DETAILED DESCRIPTION:
The investigators will identify randomised controlled trials without language restriction that meet the inclusion criteria by searching the Cochrane database, Ovid Medline, Google Scholar and other sources. The investigators will exclude observational studies, short-term trials <2 months duration, studies in pregnant diabetic subjects, newly diagnosed type 2 diabetes, trials in type 1 diabetes and extensions of previous studies.

Data on individual participants will be obtained directly from trialists and from funding sponsors who hold the trial data and will include age, sex, duration of diabetes, treatment group, baseline and final HbA1c, baseline and final insulin dose, baseline and final BMI.

A 'two-step' meta-analysis will be performed to estimate overall mean differences in HbA1c, insulin dose and weight/BMI for the trials. Then, a 'one-step' meta-regression analysis will be conducted by creating a single large dataset from the individual patient data. Determinants of final HbA1c, BMI/weight and insulin dose will be explored using Bayesian approaches with covariates that include baseline HbA1c, age, diabetes duration, BMI, insulin dose and interactions between the covariates.

ELIGIBILITY:
Inclusion Criteria:

* RCTs of CSII vs. MDI in type 2 diabetes, study duration at least 2 months, non-pregnant

Exclusion Criteria:

* Type 1 diabetes, studies <2 months duration, pregnant women, newly diagnosed type 2 diabetes and extensions of previous studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | Up to 24 months
  Difference in glycaemic control between treatments, as measured by HbA1c

SECONDARY OUTCOMES:
Insulin dose | Up to 24 months
  Difference in insulin dose between treatments
Weight or BMI | Up to 24 months
  Difference in weight or BMI between treatments

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Pickup JC, Reznik Y, Sutton AJ. Glycemic Control During Continuous Subcutaneous Insulin Infusion Versus Multiple Daily Insulin Injections in Type 2 Diabetes: Individual Patient Data Meta-analysis and Meta-regression of Randomized Controlled Trials. Diabetes Care. 2017 May;40(5):715-722. doi: 10.2337/dc16-2201. PMID 28428322